CLINICAL TRIAL: NCT01866046
Title: Rapid HIV Testing and Counseling in High Risk Women in Shelters
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Akron (Other)
Collaborators: Brown University (Other); The Miriam Hospital (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Dawn Johnson, Associate Professor, The University of Akron
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21NR013628-02 (NIH)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: HIV Risk
Keywords: battered women; HIV risk; STI risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RESPECT-IPV (Experimental): Rapid HIV testing and risk prevention intervention for victims of intimate partner violence
  Interventions: Behavioral: RESPECT-IPV

INTERVENTIONS:
Behavioral: RESPECT-IPV — rapid HIV testing intervention and behavioral counseling session where identify risks and develop a risk reduction plan

SUMMARY:
This is a developmental study evaluating a new rapid HIV testing and risk prevention intervention for residents of battered women's shelters who endorse risky sexual behaviors.

DETAILED DESCRIPTION:
A. Specific Aims More than one million Americans are living with HIV, with over 20% unaware of their HIV status. Early detection of HIV status is crucial to prevent transmission to others and to link those who are HIV positive to medical care and other clinical services. Consistently, the National HIV/AIDS strategy has established a goal of increasing the awareness of HIV status in Americans from 79% to 90% within the next four years. Thus, there is a strong need for increased testing efforts, particularly among high risk, underserved populations. To be effective, these testing efforts need to address many of the barriers to testing and linkage to care faced by these underserved populations. Victims of intimate partner violence (IPV) are one such underserved population who are at high risk for HIV infection and face many barriers to testing and linkage to care.

IPV is a pervasive public health problem with 25% of women reporting IPV in their lifetime. A growing body of literature highlights the association between IPV and HIV risk. IPV victims are more likely to engage in HIV risk behaviors, including unprotected sex, sex with risky partners (e.g., HIV-positive, injection drug users), sex with more than one sex partner, and trading sex, and are more likely to have a sexually transmitted disease (STI). Additionally, posttraumatic stress disorder (PTSD) and substance use disorder (SUD), highly prevalent in IPV victims, are associated with high risk sexual behaviors. Furthermore, women with IPV underutilize medical care and often encounter numerous barriers to health care (e.g., transportation, under or un-insured). Unfortunately, very few HIV prevention interventions have been developed or tested for this vulnerable and underserved population of women.

IPV Victims in domestic shelters are at significant risk for HIV (i.e., 69-87% report unprotected sex and 33% report having an STI). Domestic violence shelters also present an opportune setting for providing health care services for women. There are approximately 2,000 community-based shelter programs throughout the US, providing emergency shelter to approximately 300,000 women and children each year. Considering the number of women who seek help from these facilities and that IPV victims who seek shelter have already instituted a change in their life, a prime time to intervene may be while these women are already seeking help from these community based organizations. Further, domestic shelters provide a safe and supportive environment which is ideal for HIV testing and prevention. Thus incorporating HIV testing and prevention within domestic shelters will provide access to a significant population of women with an overall high risk for HIV infection while significantly reducing many of the barriers to testing and linkage to care faced by IPV victims. Rapid HIV testing allows for provision of HIV testing, counseling, and test results in one visit, eliminating the problem of clients not returning for test results. Thus, rapid testing offers an ideal option for residents of domestic shelters, given their multiple competing demands and barriers to traditional HIV testing and prevention. RESPECT is an evidence-based CDC Diffusion of Effective Behavioral Interventions (DEBI), utilizing a client-focused, interactive HIV risk reduction counseling model delivered in conjunction with HIV testing. RESPECT-2, which has been adapted for use with rapid testing, is brief and easily adaptable to many clinical settings. IPV victims, however, face distinct HIV risk factors, such as difficulty in negotiating condom use and other preventative sexual behaviors, out of fear of retaliation or being raped by their abusive partner. Hence, RESPECT-2 needs to be tailored to meet the specific needs of our target population.

The Specific Aims of this R21 Exploratory/Developmental Research Proposal are to (a) expand RESPECT-2 for our target population (i.e., RESPECT-IPV) and (b) to collect preliminary data on RESPECT-IPV + rapid testing's feasibility, acceptability, and initial efficacy in residents of domestic shelters. To facilitate sustainability and future dissemination of RESPECT-IPV + rapid testing, the intervention will be delivered by trained personnel from community-based CDC supported counseling, testing, and referral (CTC) sites.

The development aim of this R21 proposal is to develop the manual for RESPECT-IPV, incorporating information gathered from four focus groups with IPV victims and two focus groups with shelter staff, the literature on IPV and HIV risk, and a pre-pilot open trial to increase acceptability of RESPECT-IPV and to tailor the intervention to meet the unique needs of our target population. The pilot study aims of this R21 proposal are to: (1) Assess the feasibility and acceptability of RESPECT-IPV + rapid testing in a sample of 100 high-risk shelter women. Predictors of acceptability (e.g., PTSD symptoms, substance use, IPV severity, prior testing history, HIV knowledge, HIV risk behavior, HIV anxiety, stage of change) will also be explored. (2) Conduct an open trial of RESPECT-IPV + rapid testing in a sample of 100 high-risk shelter women and examine preliminary evidence for the hypotheses that RESPECT-IPV will be associated with reduced unprotected vaginal or anal sex occasions (USOs) at 1-week and 3-months after leaving shelter and fewer cases of vaginal trichomoniasis 3-months after leaving shelter. Secondary outcomes include HIV knowledge, risk intentions, and other HIV risk behaviors (e.g. multiple partners, substance use). As a result we will have created a novel testing and counseling intervention for high-risk, underserved, shelter women, providing the groundwork to test RESPECT-IPV's efficacy in future R01 clinical trials and dissemination studies.

ELIGIBILITY:
Inclusion Criteria:

* intimate partner violence and at least one unprotected sexual occasion 3 months prior to entering shelter

Exclusion Criteria:

* HIV positive

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
number of unprotected sexual occasions | up to 3 months post shelter
  Calendar assessment of number of unprotected sexual occasions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Akron, Akron, Ohio, United States

REFERENCES:
- [Derived] Johnson DM, Johnson NL, Beckwith CG, Palmieri PA, Zlotnick C. Rapid Human Immunodeficiency Virus Testing and Risk Prevention in Residents of Battered Women's Shelters. Womens Health Issues. 2017 Jan-Feb;27(1):36-42. doi: 10.1016/j.whi.2016.10.007. Epub 2016 Nov 30. PMID 27914861